CLINICAL TRIAL: NCT04188912
Title: Close Assessment and Testing for Chronic GVHD (The CATCH Study)
Brief Title: Close Assessment and Testing for Chronic Graft Versus Host Disease, CATCH Study
Acronym: CATCH
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: RG1005155; NCI-2019-07293 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10134 (Other: Fred Hutch/University of Washington Cancer Consortium); U01CA236229 (NIH)
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue, saliva, tears, buccal mucosa, feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (sample collection, survey, imaging, spirometry): Patients undergo collection of tears, saliva, buccal mucosa, and fecal samples before stem cell transplant, at 2-3, 4, 6, 8, 10, and 12 months after stem cell transplant, and at cGVHD onset. Patients also undergo collection of blood samples before stem cell transplant, at 1-2, 2-3, 4, 6, 8, 10, and 12 months after stem cell transplant, and at cGVHD onset. Patients may undergo skin and mouth biopsy over 15-30 minutes before stem cell transplant, at 2-3 and 12 months after stem cell transplant, and at cGVHD onset. Patients undergo digital pictures of the eyes, mouth and skin, and optical coherence tomography before stem cell transplant, at 2-3, 4, 6, 8, 10, and 12 months after stem cell transplant, and at cGVHD onset. Patients without standard of care formal pulmonary function test undergo portable spirometry at 2-3, 4, 6, 8, 10, and 12 months after stem cell transplant, and at cGVHD onset. Patients also complete surveys and have their medical records reviewed.
  Interventions: Procedure: Biospecimen Collection; Procedure: Optical Coherence Tomography; Procedure: Spirometry; Other: Survey Administration; Other: Digital Photography; Other: Quality-of-Life Assessment; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, tears, saliva, buccal mucosa, feces, and tissue samples
Procedure: Optical Coherence Tomography — Undergo optical coherence tomography
  Other Names: OCT
Procedure: Spirometry — Undergo portable spirometry
Other: Survey Administration — Complete survey
Other: Digital Photography — Undergo digital photography
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Medical Chart Review — Review of medical charts
  Other Names: Chart Review

SUMMARY:
This trial observes and collects samples from patients before and after stem cell transplantation to learn more about how and why a complication called chronic graft-versus-host disease (GVHD) develops after stem cell transplantation. Performing close observation and various types of testing may enable doctors to notice symptoms or problems sooner than they would normally have been noticed and predict which patients will develop chronic GVHD.

DETAILED DESCRIPTION:
OUTLINE:

Patients undergo collection of tears, saliva, buccal mucosa, and fecal samples before stem cell transplant, at 2-3, 4, 6, 8, 10, and 12 months after stem cell transplant, and at cGVHD onset. Patients also undergo collection of blood samples before stem cell transplant, at 1-2, 2-3, 4, 6, 8, 10, and 12 months after stem cell transplant, and at cGVHD onset. Patients may undergo skin and mouth biopsy over 15-30 minutes before stem cell transplant, at 2-3 and 12 months after stem cell transplant, and at cGVHD onset. Patients undergo digital pictures of the eyes, mouth and skin, and optical coherence tomographybefore stem cell transplant, at 2-3, 4, 6, 8, 10, and 12 months after stem cell transplant, and at cGVHD onset. Patients without standard of care formal pulmonary function test undergo portable spirometry at 2-3, 4, 6, 8, 10, and 12 months after stem cell transplant, and at cGVHD onset. Patients also complete surveys and have their medical records reviewed.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older
* Scheduled for allogeneic HCT from any donor for any indication, with a risk of cGVHD of > 25% (see below in exclusion criteria for treatment plans with a cGVHD risk < 25%)
* Ability and willingness to comply with the intensive assessment schedule including evaluation every other month at a participating site
* Ability to communicate in English or Spanish, to allow completion of patient surveys and clear communication with the study team

Exclusion Criteria:

* Receipt of umbilical cord blood, bone marrow with post-transplant cyclophosphamide (peripheral blood with post-transplant cyclophosphamide is allowed), anti-thymocyte globulin, alemtuzumab, or ex-vivo T-cell depletion. These patients are excluded because they have a cGVHD risk of < 25%
* Hematologic malignancy with active disease at the time of transplant. Minimal residual disease is allowed
* Hematopoietic cell transplant co-morbidity index > 4 based on parameters known at time of enrollment
* Prior allogeneic transplant
* Prior autoimmune disease with ongoing symptoms
* History of noncompliance
* Inability to comply with study requirements due to geographic, logistic, social or any other factors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for allogeneic hematopoietic cell transplantation (HCT) from any donor for any indication, with a risk of cGVHD of > 25%
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Levels of cytokines | Up to 3 years
  Will compare the pg/ml levels and trajectories of proteins (IL-1b; IL-4; IL-5; IL-6; IL-8; IL-10; IL-13; IL-17a (pg/mL); TNF; G-CSF; IFNgamma; MCP-1; IL-12p40; GM-CSF; IL-2) between patients who do and do not develop chronic graft versus host disease (cGVHD). Blood will be analyzed separately from saliva and conjunctival washings.
Onset of cGVHD | Up to 3 years
  Onset of cGVHD will be treated as a time-to-event endpoint, using Cox regression with monthly levels or slopes of the markers entered as time dependent covariates.
Percentage of cellular populations | Up to 3 years
  Will compare the levels, proportions and trajectories of different cellular populations between those with and without cGVHD, and with different cGVHD organ involvement and symptoms. The following cell subtypes are of highest interest: Th17, FOXP3+ T regulatory cells, FOXP3- T regulatory type 1 (TR1) cells, T follicular helper cells, activated B cells, B regulatory cells, and monocytes but the list may evolve before actual testing.
Number of patients with tissue alterations in skin, mouth and eyes | Up to 3 years
  Tissue alterations will be classified into Abnormal and Normal, and measured by biopsy and/or advanced bioimaging techniques. Histologic findings, ribonucleic acid (RNA) expression profiles, optical coherence tomography (OCT) findings and digital image interpretations will be compared between patients who do and do not develop cGVHD or who have different cGVHD clinical phenotypes and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (7):
- United States (7):
  - University of Florida, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - National Cancer Institute, Bethesda, Maryland
  - Roswell Park, Buffalo, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt, Nashville, Tennessee
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pidala J, Carpenter PA, Onstad L, Pavletic SZ, Hamilton BK, Chen GL, Farhadfar N, Hall M, Lee SJ. Study protocol: Close Assessment and Testing for Chronic Graft-vs.-Host disease (CATCH). PLoS One. 2024 May 16;19(5):e0298026. doi: 10.1371/journal.pone.0298026. eCollection 2024. PMID 38753616